CLINICAL TRIAL: NCT03179137
Title: Pathophysiological Mechanisms Elicited by Ischemia and Metabolic Co-morbidities in Myocardium of Patients With Coronary Artery Disease
Brief Title: Mitochondrial Bioenergetics and Role in Cellular Damage in Ischemic Myocardium
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2181-198-03
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus; Mitochondrial Metabolism Disorders
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human myocardial tissue, atrial and ventricular; Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard therapy — Patients with therapy prescribed independent of the study

SUMMARY:
Cardiac ischemia is a common pathological condition, known to elicit multiple pathological processes at the cellular level. One of the most affected is thought to be cellular metabolism, key for the adequate cardiac function. The aim is to study mitochondrial bioenergetic function, interaction with other cellular systems and influence of several co-morbidities in myocardium of the affected patients.

DETAILED DESCRIPTION:
Coronary artery disease, one of the most common pathologies in the developed world, causes hypoperfusion of myocardial tissue, usually evident by the presence of anginal pain. This myocardial ischemia elicits alterations in normal cardiomyocyte physiology, which gradually deteriorate cellular function, affecting the performance of the entire organ. The condition is frequently further complicated (and aggravated) by the presence of various co-morbidities, such as diabetes mellitus. The primary aim of this study is to investigate the cardiomyocyte bioenergetics and the consequences of potentially reduced mitochondrial metabolic function in ischemic heart, and evaluate the potential contribution of other conditions, primarily ones affecting metabolic homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease
* Indication for coronary artery bypass grafting surgery

Exclusion Criteria:

* Emergency patients
* Patients with LV ejection fraction (LVEF) below 30%
* Patients with severe renal, hepatic or pulmonary disease

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodynamically stable patients with coronary artery disease diagnosed with angiography with indication for coronary artery bypass grafting surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial oxygen consumption (rate of oxygen consumption per milligram of left ventricular tissue) | 2016-2020
  Mitochondrial respiration in nmol O2/minute/mg of tissue weight will be measured as an indicator of mitochondrial ATP production capacity, using different metabolic substrates
Myocardial production of reactive oxygen species | 2016-2020
  Myocardial production of reactive oxygen species will be measured using electron paramagnetic resonance and fluorometry

SECONDARY OUTCOMES:
Anti-cardiolipin antibodies in the blood of patients with symptoms of cardiac ischemia | 2016-2020
  Anticardiolipin antibodies assessed in venous blood of patients with angina pectoris undergoing coronary angiography

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, University of Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03179137/Prot_000.pdf